CLINICAL TRIAL: NCT00691002
Title: Calcipotriol Plus Hydrocortisone in Psoriasis Vulgaris on the Face and on the Intertriginous Areas
Brief Title: Efficacy and Safety of Calcipotriol Plus Hydrocortisone Ointment in Psoriasis Vulgaris on the Face and Skin Folds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEO 80190-O21
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2021-08-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2021-08

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LEO 80190 (Experimental): Calcipotriol 25 mcg/g plus 10 mg/g hydrocortisone ointment (LEO 80190)
  Interventions: Drug: Calcipotriol plus hydrocortisone (LEO 80190)
- LEO 80190 vehicle (Placebo Comparator): Ointment Vehicle
  Interventions: Drug: LEO 80190 Vehicle
- Calcipotriol (Active Comparator): Calcipotriol 25 mcg/g in the ointment vehicle
  Interventions: Drug: Calcipotriol
- Hydrocortisone (Active Comparator): Hydrocortisone 10 mg/g in the ointment vehicle
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Calcipotriol plus hydrocortisone (LEO 80190) — Once daily application
  Arms: LEO 80190
Drug: LEO 80190 Vehicle
  Arms: LEO 80190 vehicle
Drug: Hydrocortisone
  Arms: Hydrocortisone
Drug: Calcipotriol
  Arms: Calcipotriol

SUMMARY:
There are few therapies suitable for the treatment of psoriasis on the face and skin folds. As these areas are sensitive, irritation and other adverse reactions are more common than elsewhere on the body. The purpose of the study is to compare the efficacy and safety of once daily treatment for up to 8 weeks of an ointment containing calcipotriol 25 mcg/g plus hydrocortisone 10 mg/g with calcipotriol 25 mcg/g in the ointment vehicle, hydrocortisone 10 mg/g in the ointment vehicle and the ointment vehicle alone in patients with psoriasis vulgaris on the face and on the intertriginous areas (= double-blind phase). Furthermore, the safety and efficacy will be evaluated for up to 60 weeks treatment as required of calcipotriol 25 mcg/g plus hydrocortisone 10 mg/g ointment in psoriasis vulgaris on the face and intertriginous areas (= open-label phase).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis vulgaris involving the face
* Clinical signs of psoriasis vulgaris on the trunk and/or the limbs, or earlier diagnosed with psoriasis vulgaris on the trunk and/or the limbs
* An extent of psoriatic involvement of the face of at least 10 cm2 (the sum of all facial lesions)
* Treatment areas (the face and the intertriginous areas) amenable to topical treatment with a maximum of 100 g of ointment per week
* Disease severity graded as mild, moderate, severe or very severe according to the investigator's global assessment of disease severity of the face

Exclusion Criteria:

* Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, vitamin D analogues, retinoids, immunosuppressants) within the 4-week period prior to randomisation
* Systemic use of biological treatments, whether marketed or not, directed against or with a potential effect on psoriasis vulgaris (e.g., alefacept, efalizumab, etanercept, infliximab, adalimumab) within 3 months prior to randomisation
* PUVA therapy or Grenz ray therapy within the 4-week period prior to randomisation
* UVB therapy within the 2-week period prior to randomisation
* Topical treatment of the face and the intertriginous areas within the 2-week period prior to randomisation (use of emollients is allowed on treatment areas during this 2-week period, but not during the double-blind phase of the study)
* Topical treatment with very potent WHO group IV corticosteroids within the 2-week period prior to randomisation
* Initiation of or expected changes in concomitant medication that may affect psoriasis vulgaris (e.g., beta blockers, anti-malaria drugs, lithium and ACE inhibitors) during the study
* Current diagnosis of erythrodermic, exfoliative, guttate or pustular psoriasis
* Patients with any of the following conditions present on the treatment area: viral (e.g., herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, perioral dermatitis, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, acne rosacea, ulcers and wounds
* Other inflammatory skin diseases (e.g., seborrhoiec dermatitis, contact dermatitis and cutaneous mycosis) that may confound the evaluation of psorisis vulgaris on the face or on the intertriginous areas
* Planned exposure to sun, UVA or UVB that may affect the psoriasis vulgaris during the study
* Known or suspected severe renal insufficiency or severe hepatic disorders
* Known or suspected disorders of calcium metabolism associated with hypercalcaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1245 (Actual)
Dates: Start 2008-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bieber, MD, Principal Investigator — Department of Dermatology and Allergy, University of Bonn
Locations (11):
- Croatia (3):
  - Croatia - managed by CRO, Zagreb
  - Macedonia - managed by CRO, Zagreb
  - Slovenia - managed by CRO, Zagreb
- Department of Dermatology and Allergy, University of Bonn, Bonn, Germany
- Poland (6):
  - Czech Republic - managed by CRO, Warsaw
  - Hungary - managed by CRO, Warsaw
  - Latvia - managed by CRO, Warsaw
  - Poland - managed by CRO, Warsaw
  - Belgium - managed by CRO, Warsaw
  - The Netherlands - managed by CRO, Warsaw
- Serbia - managed by CRO, New Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1245 subjects were enrolled (informed consent signed and CRF started). Five subjects left the study during washout (2 screening failures, 2 lost to follow-up and 1 unacceptable adverse event). One subject attended Visit 1 but was not randomized (voluntary withdrawal). Therefore, 1239 of the enrolled subjects were randomized in the study.
Pre-assignment Details: The Randomized double-blind phase of the study lasted up to 8 weeks, and was followed by a 52-week Open-label period in which participants had the opportunity to receive Calcipotriol 25 mcg/g plus 10 mg/g Hydrocortisone ointment.
Groups:
- LEO 80190: Once daily application Calcipotriol 25 mcg/g plus 10 mg/g hydrocortisone ointment (LEO 80190)
- Calcipotriol: Once daily application
  Calcipotriol 25 mcg/g in the ointment vehicle
- Hydrocortisone: Once daily application
  Hydrocortisone 10 mg/g in the ointment vehicle
- LEO 80190 Vehicle: Once daily application
  Ointment Vehicle
- Open-label Phase: LEO 80190 ointment : calcipotriol 25 mcg/g plus 10 mg/g hydrocortisone ointment
Period: 8-week, Double-blind, 4-arm
Arm/Group | LEO 80190 | Calcipotriol | Hydrocortisone | LEO 80190 Vehicle | Open-label Phase
Started | 353 | 342 | 363 | 181 | 0
Completed | 325 | 308 | 340 | 169 | 0
Not Completed | 28 | 34 | 23 | 12 | 0
Period: 52-week, Open-label, Single Arm
Arm/Group | LEO 80190 | Calcipotriol | Hydrocortisone | LEO 80190 Vehicle | Open-label Phase
Started | 454 | 0 | 0 | 0 | 0
Completed | 403 | 0 | 0 | 0 | 0
Not Completed | 51 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 80190 | Calcipotriol | Hydrocortisone | LEO 80190 Vehicle | Total
Number analyzed (Participants) | 353 | 342 | 363 | 181 | 1239
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (15.3) | 44.8 (15.1) | 43.0 (14.1) | 44.6 (15.1) | 43.6 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 139 | 147 | 76 | 517
  Male | 198 | 203 | 216 | 105 | 722
Region of Enrollment [Number; unit: participants]
  Belgium | 4 | 6 | 5 | 2 | 17
  Croatia | 15 | 13 | 16 | 7 | 51
  Czechia | 29 | 22 | 24 | 15 | 90
  Germany | 99 | 95 | 96 | 55 | 345
  Hungary | 58 | 59 | 64 | 35 | 216
  Latvia | 23 | 20 | 24 | 10 | 77
  Macedonia | 7 | 8 | 8 | 3 | 26
  Netherlands | 4 | 6 | 5 | 1 | 16
  Poland | 79 | 76 | 80 | 37 | 272
  Serbia | 34 | 36 | 40 | 16 | 126
  Slovenia | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Participants With "Controlled Disease" According to the Investigator's Global Assessment(IGA) of Disease Severity of the Face at Week 8 (Visit 6) in the Double-blind Phase
Description: The (sub) investigator made an assessment of the disease severity of the face using the 6-category scale below.
  Clear, Almost clear, Mild, Moderate, Severe, Very severe
  The assessment was made considering the condition of psoriasis vulgaris of the face at the time of the evaluation, not in relation to the condition at a previous visit.
  For subjects with a baseline (Visit 1) severity of moderate or worse - "controlled disease" of the face was defined as clear or almost clear according to the IGA of disease severity of the face.
  For subjects with a baseline (Visit 1) severity of mild - "controlled disease" of the face was defined as clear according to the IGA of disease severity of the face.
Time Frame: At Week 8 (end of treatment for double-blind phase)
Measure: Count of Participants; unit: Participants
Groups:
- LEO 80190: Once daily application Calcipotriol plus hydrocortisone (LEO 80190)
Arm/Group | LEO 80190 | Calcipotriol | Hydrocortisone | LEO 80190 Vehicle
Number analyzed (Participants) | 353 | 341 | 363 | 180
Participants | 158 | 135 | 115 | 41
Statistical Analysis 1: Comparison: LEO 80190 vs Calcipotriol; Test for superiority of LEO 80190 ointment versus calcipotriol ointment at Week 8 LOCF (Last Observation Carried Forward); Test type: Superiority; p = 0.11, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.94 to 1.74]
Statistical Analysis 2: Comparison: LEO 80190 vs Hydrocortisone; Test for superiority of LEO 80190 ointment versus hydrocortisone ointment at Week 8 LOCF (Last Observation Carried Forward); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.31 to 2.45]
Statistical Analysis 3: Comparison: LEO 80190 vs LEO 80190 Vehicle; Test for superiority of LEO 80190 ointment versus ointment vehicle at Week 8 LOCF (Last Observation Carried Forward); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.70, 95% CI 2-sided [1.80 to 4.04]

2. Secondary Outcome: Participants With "Controlled Disease" According to the IGA of Disease Severity of the Face at Week 4 (Visit 4) in the Double-blind Phase
Description: The assessment of the disease severity of the face was made using the 6-category scale below.
  Clear Almost clear Mild Moderate Severe Very severe
  The assessment was made considering the condition of psoriasis vulgaris of the face at the time of the evaluation, not in relation to the condition at a previous visit.
  For subjects with a baseline severity of moderate or worse - "controlled disease" of the face was defined as clear or almost clear according to the IGA of disease severity of the face.
  For subjects with a baseline severity of mild - "controlled disease" of the face was defined as clear according to the IGA of disease severity of the face.
Time Frame: At Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80190 | Calcipotriol | Hydrocortisone | LEO 80190 Vehicle
Number analyzed (Participants) | 353 | 341 | 363 | 180
Participants | 101 | 66 | 61 | 14

3. Secondary Outcome: Participants With "Success" According to Total Sign Score (TSS) of the Face at Week 8 (Visit 6) in the Double-blind Phase
Description: "Success" was defined as a TSS score of 0 or 1.
  For each clinical sign, a single score, reflecting the average severity of all psoriatic lesions on the face was determined according to the scale below:
  Redness 0 = none (no erythema) 1 = mild (faint erythema, pink to very light red) 2 = moderate (definite light red erythema) 3 = severe (dark red erythema) 4 = very severe (very dark red erythema) Thickness 0 = none (no plaque elevation) 1 = mild (slight, barely perceptible elevation) 2 = moderate (definite elevation but not thick) 3 = severe (definite elevation, thick plaque with sharp edge) 4 = very severe (very thick plaque with sharp edge) Scaliness 0 = none (no scaling) 1 = mild (sparse, fine-scale lesions, only partially covered) 2 = moderate (coarser scales, most of lesions covered) 3 = severe (entire lesion covered with coarse scales) 4 = very severe (very thick coarse scales, possibly fissured)
  The sum of the three scores constituted a TSS ranging from 0 to 12
Time Frame: At Week 8 (end of treatment for double-blind phase)
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80190 | Calcipotriol | Hydrocortisone | LEO 80190 Vehicle
Number analyzed (Participants) | 353 | 341 | 363 | 180
Participants | 171 | 136 | 131 | 42

4. Secondary Outcome: Participants With "Controlled Disease" According to the IGA of Disease Severity of the Intertriginous Areas at Week 8 (Visit 6) in the Double-blind Phase
Description: The (sub)investigator made an assessment of the disease severity of the intertriginous areas using the 6-category scale below.
  Clear, Almost clear, Mild, Moderate, Severe, Very severe The assessment was made considering the condition of psoriasis vulgaris of the intertrigi-nous areas at the time of the evaluation, not in relation to the condition at a previous visit.
  For subjects with a baseline severity of moderate or worse - "controlled disease" of the intertriginous areas was defined as clear or almost clear according to the IGA of disease severity of the intertriginous areas.
  For subjects with a baseline severity of mild - "controlled disease" of the intertriginous areas was defined as clear according to the IGA of disease severity of the intertriginous areas.
Time Frame: At Week 8 (end of treatment for double-blind phase)
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80190 | Calcipotriol | Hydrocortisone | LEO 80190 Vehicle
Number analyzed (Participants) | 171 | 173 | 182 | 89
Participants | 80 | 55 | 48 | 14

5. Secondary Outcome: Participants With "Success" According to Total Sign Score of the Intertriginous Areas at Week 8 (Visit 6) in the Double-blind Phase
Description: The severity of the subject's psoriasis vulgaris on the intertriginous areas was evaluated in terms of the three clinical signs: redness, thickness and scaliness. All the defined intertriginous areas were rated separately using the same scale as for the investigator's assessment of clinical signs (redness, thickness and scaliness) of the face.
  For each clinical sign, a single score, reflecting the average severity of all psoriatic lesions on the face was determined according to the scale below:
  Redness 0 = none
  1. = mild
  2. = moderate
  3. = severe
  4. = very severe
  Thickness 0 = none
  1. = mild
  2. = moderate
  3. = severe
  4. = very severe
  Scaliness 0 = none
  1. = mild
  2. = moderate
  3. = severe
  4. = very severe
  A mean score was calculated for each sign (redness, thickness and scaliness) based on scores of all the defined intertriginous areas with psoriasis at baseline and the sum of these mean scores constituted the TSS.
  "Success" was defined as a TSS score of 0 or 1.
Time Frame: At Week 8 (end of treatment for double-blind phase)
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80190 | Calcipotriol | Hydrocortisone | LEO 80190 Vehicle
Number analyzed (Participants) | 171 | 173 | 182 | 89
Participants | 82 | 81 | 59 | 15

ADVERSE EVENTS:
Time Frame: Double-blind Phase: From baseline (Day 0) to end of trial (Day 56±2) + Follow-up (Day 14±2) Open-label Phase: From Week 8 to Week 60 ±7 days + Follow-up (Day 14±2)
Description: The adverse events where collected for the the safety analysis set (SAS). The SAS consisted of those randomized patients who received any treatment with trial medication and for whom the presence or confirmed absence of adverse events were available. In total, 1235 subjects are included in the safety analysis set.
Arm/Group | LEO 80190 | Calcipotriol | Hydrocortisone | LEO 80190 Vehicle | Open-label Phase
All-Cause Mortality (participants affected / at risk) | 0/351 | 0/341 | 0/362 | 0/181 | 0/453
Serious Adverse Events (participants affected / at risk) | 5/351 | 5/341 | 4/362 | 0/181 | 24/453
Other Adverse Events (participants affected / at risk) | 91/351 | 100/341 | 70/362 | 47/181 | 266/453
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 80190 (N=351) | Calcipotriol (N=341) | Hydrocortisone (N=362) | LEO 80190 Vehicle (N=181) | Open-label Phase (N=453)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Deafness traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cervical vertebra injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 2
Panic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Knee operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 80190 (N=351) | Calcipotriol (N=341) | Hydrocortisone (N=362) | LEO 80190 Vehicle (N=181) | Open-label Phase (N=453)
Diarrhoea (Gastrointestinal disorders) | 4 | 6 | 0 | 0 | 9
Toothache (Gastrointestinal disorders) | 4 | 1 | 1 | 0 | 5
Application site pruritus (General disorders) | 2 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 4 | 2 | 3 | 2 | 9
Herpes simplex (Infections and infestations) | 4 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 3 | 2 | 2 | 2 | 10
Nasopharyngitis (Infections and infestations) | 8 | 5 | 12 | 11 | 55
Burning sensation (Nervous system disorders) | 5 | 12 | 1 | 4 | 0
Headache (Nervous system disorders) | 11 | 6 | 8 | 2 | 17
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 4 | 0 | 13
Erythema (Skin and subcutaneous tissue disorders) | 7 | 24 | 7 | 7 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 14 | 3 | 5 | 8
Psoriasis (Skin and subcutaneous tissue disorders) | 26 | 23 | 27 | 12 | 114
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 6
Cystitis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 5
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 9
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 6
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 10
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 8
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Company acknowledges the investigators' right to publish the entire results of the study, irrespective of outcome. The Company retains the right to have any publication submitted to the Company for review at least 30 days prior to the same paper being submit-ted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.